CLINICAL TRIAL: NCT00040508
Title: Sirolimus for Focal Segmental Glomerulosclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 020235; 02-DK-0235
Record Dates: First submitted 2002-06-26; First posted 2002-06-27 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-01

CONDITIONS: Focal Glomerulosclerosis
Keywords: Proteinuria; Renal Failure; Fibrosis; Rapamycin; Immunosuppression; Focal Segmental Glomerulosclerosis; FSGS
MeSH Terms: conditions — Glomerulosclerosis, Focal Segmental; Proteinuria; Renal Insufficiency; Fibrosis | interventions — Sirolimus

INTERVENTIONS:
Drug: Sirolimus

SUMMARY:
This study will determine the safety and effectiveness of sirolimus (Rapamune® (Registered Trademark)) in treating focal segmental glomerulosclerosis (FSGS), a disease involving kidney scarring and increased protein in the urine. About one-half of patients with FSGS go on to develop end-stage kidney disease within 6 years, requiring dialysis or kidney transplant. Therapies to reduce urine protein are likely to stop the progression of renal scarring and reduce the chance of developing kidney failure. However, current treatments for FSGS, such as prednisone, cyclophosphamide, and cyclosporine, are not effective in many patients and can cause serious side effects. This study will see if sirolimus, a drug with both anti-scarring and immune suppressing properties, can lower the amount of protein in the urine and slow or stop the kidney disease.

Patients 13 years of age and older with FSGS who have had at least one standard treatment for FSGS may be eligible for this 24-month study. Pregnant and nursing women may not participate. Candidates will be screened with a medical history and physical examination, review of medical records and kidney biopsy, 24-hour urine collection, and blood tests.

Participants will take sirolimus tablets once a day for 1 year. Three 24-hour urine collections will be done before starting treatment. Blood will be drawn to measure drug levels every week for the first month after starting treatment, then every other week for 1 month, and then every 2 months until treatment stops. Patients who do not have a complete response to the drug at low levels will have their dose increased. Patients will be seen at the NIH clinic in Bethesda, Md., for the screening visit and then at 1, 4, 8, 12, and 15 months for blood and urine tests. Additional urine collections and blood tests will be done periodically throughout the 24-month study period by the patient's local physician.

Patients whose urine protein decreases on therapy will be asked to wait 3 months before starting another treatment and will monitored during that time to determine if the response is sustained. Patients whose urine protein levels do not decrease with sirolimus will not be asked to wait 3 months before starting another therapy. Follow-up with the local physician will continue at 18 and 24 months after starting the study.

Patients whose urine protein levels increase with sirolimus treatment will be taken off the study and may seek other treatment at any time.

DETAILED DESCRIPTION:
Sirolimus is an immunosuppressive agent that was recently approved for use in organ transplantation. We propose to carry out a pilot study whose objectives are to determine the safety and efficacy profile of sirolimus in focal segmental glomerulosclerosis (FSGS). Current therapy for FSGS has limited efficacy. Sirolimus was selected for the following reasons: 1) sirolimus reduces proliferation of mesangial cells and endothelial cells, 2) sirolimus reduces fibrosis in experimental models of liver and kidney disease, 3) sirolimus is a potent immunosuppressive, and other immunosuppressives including glucocorticoids and cyclosporine have shown some efficacy in FSGS, and 4) sirolimus may have a direct anti-proteinuric effect, as suggested by in vitro studies. We will recruit up to 30 patients, including adults and children greater than or equal to 13.0 years of age. The study design is open label, with therapy for one year using doses adjusted to achieve trough levels of 5-15 ng/mL during the first 4 months and if a complete remission is not achieved and sustained, 10-20 ng/mL during the remainder of the study. The primary outcome will be reduction in proteinuria, categorized as complete remission and partial remission, comparing baseline values and 12 month values. The study will recruit patients in two groups: 1) a drug washout group, for patients who can tolerate receiving no immunosuppressive therapy for 4 weeks prior to initiating sirolimus therapy, and 2) a drug overlap group, for patients who cannot tolerate cessation of immunosuppressive therapy due to severe edema or other complications of nephrotic syndrome; these patients will receive prednisone for up to 6 months while taking sirolimus (with a target of prednisone less than 20 mg QOD by month 3) or will receive cyclosporine, tacrolimus, or mycophenolate mofetil for up to 4 weeks while initiating sirolimus therapy.

ELIGIBILITY:
INCLUSION CRITERIA

Renal biopsy showing FSGS, including all variants with the exception of HIV-associated FSGS.

Nephrotic range proteinuria, defined as 24 hour urine protein excretion greater than or equal to 3.5 g/d in adults and children weighing greater than or equal to 70 kg and greater than or equal to 50 mg/kg in adults or children weighing less than 70 kg. Proteinuria will be assessed with at least three 24 hour urine collections obtained during the baseline period (for these collections, there is no minimum period, the maximum period is 3 months prior to study entry, and the most recent must be within 1 month of entry). These measurements will be obtained while on angiotensin antagonist therapy (if tolerant of this medication) and will exclude urine collections judged inadequate based on creatinine appearance. For patients in the drug overlap group, baseline proteinuria will be determined from patient's records demonstrating on at least one urine collection, proteinuria greater than 3.5 g/d while off immunosuppressive therapy.

Ability and willingness to provide informed consent (adults greater than or equal to 18.0 years) or assent (children greater than or equal to 13.0 years).

Completion of a therapeutic trial of at least one of the following, without sustained CR:

Steroid therapy for greater than or equal to 8 weeks, either daily or alternate day or intermittent (oral or parenteral)

Cyclosporine or tacrolimus or mycophenolate mofetil for greater than or equal to 3 months

Cyclophosphamide (either oral or intravenous) or chlorambucil for greater than or equal to three months

EXCLUSION CRITERIA

Intolerance to sirolimus or prior use of sirolimus for FSGS.

Estimated GFR less than 30 mL/min/1.73m(2). The rational is that 1) sirolimus therapy is most likely to be beneficial during the early phase of FSGS, before progressive fibrosis in the glomeruli and interstitium has become the dominant abnormality and may be irreversible, and 2) we wish to enroll patients who are unlikely to progress to ESRD within the one year treatment period.

Patients following renal transplant. We wish to rest sirolimus with a minimum of other immunosuppressive therapy.

Children less than 13.0 years.

Uncontrolled hypertension, defined as BP greater than 140/90 on greater than 25% of measurements.

Pregnancy, lactation, or unwillingness or inability to practice effective contraception. The rationale is that the safety of sirolimus in pregnancy has not been determined and excretion via breast milk may alter pharmacokinetics.

Chronic active infections requiring treatment, including untreated reactive PPD, or any infection sufficiently severe require parenteral antibiotics during the preceding 30 days. The rationale is that immunosuppression may exacerbate infection.

HIV-1 infection or hepatitis B infection or hepatitis C infection (defined as detectable RNA off anti-viral therapy). The rationale is that immunosuppression may exacerbate infection.

Chronic liver disease sufficiently severe to impair sirolimus metabolism; this would include prolonged pro-thrombin time.

Basal thrombocytopenia less than 100,000 cells/microliter or absolute neutrophil count less than 2000 cells/microliter or hematocrit less than 30. The rationale is that sirolimus may further lower cell counts.

Cancer diagnosis or cancer recurrence within the preceding 5 years, excluding basal cell carcinoma of the skin. The rationale is that cancer progression may be accelerated by immunosuppression.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30
Dates: Start 2002-06; Study Completion 2005-01

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK), Bethesda, Maryland, United States

REFERENCES:
- [Background] Levey AS, Bosch JP, Lewis JB, Greene T, Rogers N, Roth D. A more accurate method to estimate glomerular filtration rate from serum creatinine: a new prediction equation. Modification of Diet in Renal Disease Study Group. Ann Intern Med. 1999 Mar 16;130(6):461-70. doi: 10.7326/0003-4819-130-6-199903160-00002. PMID 10075613
- [Background] Schiffmann R, Kopp JB, Austin HA 3rd, Sabnis S, Moore DF, Weibel T, Balow JE, Brady RO. Enzyme replacement therapy in Fabry disease: a randomized controlled trial. JAMA. 2001 Jun 6;285(21):2743-9. doi: 10.1001/jama.285.21.2743. PMID 11386930
- [Background] Korbet SM. Management of idiopathic nephrosis in adults, including steroid-resistant nephrosis. Curr Opin Nephrol Hypertens. 1995 Mar;4(2):169-76. doi: 10.1097/00041552-199503000-00010. PMID 7600048